CLINICAL TRIAL: NCT03335540
Title: ADaptiVe Biomarker Trial That InformS Evolution of Therapy
Brief Title: An Adaptive Study to Match Patients With Solid Tumors to Various Immunotherapy Combinations Based Upon a Broad Biomarker Assessment
Acronym: ADVISE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA028-001
Record Dates: First submitted 2017-11-06; First posted 2017-11-07 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Nivolumab; relatlimab; cabiralizumab; Ipilimumab; IDO-1 inhibitor LY3381916; linrodostat; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm B (Experimental): Combination therapy determined by biomarker assessment
  Interventions: Biological: Nivolumab; Biological: Relatlimab
- Arm C (Experimental): Combination therapy determined by biomarker assessment
  Interventions: Biological: Nivolumab; Biological: Cabiralizumab
- Arm D (Experimental): Combination therapy determined by biomarker assessment
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Arm F (Experimental): Combination therapy determined by biomarker assessment
  Interventions: Biological: Nivolumab; Drug: IDO1 Inhibitor
- Arm G (Experimental): Combination therapy determined by biomarker assessment
  Interventions: Biological: Nivolumab; Radiation: Radiation Therapy

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified day
  Other Names: BMS-936558
Biological: Relatlimab — Specified dose on specified day
  Other Names: BMS-986016
  Arms: Arm B
Biological: Cabiralizumab — Specified dose on specified day
  Other Names: BMS-986227; FPA008
  Arms: Arm C
Biological: Ipilimumab — Specified dose on specified day
  Other Names: BMS-734016
  Arms: Arm D
Drug: IDO1 Inhibitor — Specified dose on specified day
  Other Names: BMS-986205
  Arms: Arm F
Radiation: Radiation Therapy — Specified dose on specified day
  Arms: Arm G

SUMMARY:
The purpose of this study is to evaluate the treatment of solid tumors with various immunotherapy combinations. The treatment will be determined based upon a broad biomarker assessment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have an ECOG performance status of less than or equal to 1
* Participants must have had prior therapy;Participants who have received adjuvant or neoadjuvant anti-PD(L)1 therapy andprogressed within 6 months of completing therapy will be considered IO refractory.
* Participants must have at least 2 lesions with measurable disease as defined by RECIST Version 1.1

Exclusion Criteria:

* Participants with suspected, known, or progressive CNS metastases, have untreated CNS metastases, or have the CNS as the only site of disease
* Participants with carcinomatous meningitis
* Participants with other active malignancy requiring concurrent intervention

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with qualified tumor biopsy specimen at baseline | Up to 28 days
  An adequate quality tumor biopsy providing sufficient information prior to choosing a combination immunotherapy/Stereotactic Body Radiation Therapy (SBRT)

SECONDARY OUTCOMES:
Percent of change from baseline in histopathologic features | Up to 4 years
Percent of change from baseline in biomarker expression patterns | Up to 4 years
Number of Adverse Events (AEs) | Up to 4 years
Number of Serious Adverse Events (SAEs) | Up to 4 years
Number of Laboratory Abnormalities | Up to 4 years
  Any laboratory test result that is clinically significant or meets the definition of an SAE, requires the participant to have study treatment discontinued, or receive specific corrective therapy
Number of Adverse Events(AEs) leadind to discontinutaion | up to 4 years
  Number of Adverse Events leadind to discontinutaion
Number of Deaths | up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- United States (4):
  - Local Institution - 0001, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Local Institution - 0002, Baltimore, Maryland
  - Local Institution - 0003, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Luke JJ, Bever K, Hodi FS, Taube J, Massey A, Yao D, Neely J, Tam R, Lee G, Gupta A, Dutta S, Szabo P, Bao R, Reilly T. Rationale and feasibility of a rapid integral biomarker program that informs immune-oncology clinical trials: the ADVISE trial. J Immunother Cancer. 2025 May 19;13(5):e011170. doi: 10.1136/jitc-2024-011170. PMID 40389374
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm